CLINICAL TRIAL: NCT04404569
Title: An Open-Label, Multi-Center, Rollover Study to Provide Continued Treatment Access for Participants Enrolled in Studies of BXQ-350
Brief Title: Continued Treatment for Participants Enrolled in Studies of BXQ-350
Acronym: ETERNITI
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Bexion Pharmaceuticals no longer has open studies in which subjects would be eligible to rollover and continue treatment under the BXQ-350.AE protocol. Therefore, no additional subjects will be enrolled in this trial.
Sponsor: Bexion Pharmaceuticals, Inc. (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BXQ-350.AE
Record Dates: First submitted 2020-05-20; First posted 2020-05-27 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Neoplasms
Keywords: High-grade Glioma; Glioblastoma; Solid Tumor
MeSH Terms: conditions — Neoplasms; Glioma; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Continued Treatment (Experimental): Subjects who have completed the required study observation period or are still on treatment upon the closure of their respective BXQ-350 clinical study, and who are judged by the Investigator to benefit from continued treatment with BXQ-350. Treatment will begin after completion of the End of Study visit of the prior BXQ-350 clinical study.
  The established safe dose of BXQ-350 from previous adult and pediatric phase 1 studies is 2.4 mg/kg and 3.2 mg/kg respectively once every 28 days (± 3 days). BXQ-350 will be administered intravenously at the same dose level and frequency the subject was receiving at the end of the prior BXQ-350 clinical study. Subjects receiving a reduced dose at the end of the prior BXQ-350 clinical study due to toxicity may continue to receive a reduced dose.
  Interventions: Drug: BXQ-350

INTERVENTIONS:
Drug: BXQ-350 — BXQ-350 is a novel anti-neoplastic therapeutic agent configured from two components: Saposin C (SapC), an expressed (human) lysosomal protein, and the phospholipid dioleoylphosphatidyl-serine (DOPS), a phospholipid located on cell membranes (clinical formulation BXQ-350). BXQ-350 is administered by intravenous (IV) infusion in 28-day cycles
  Other Names: SapC-DOPS

SUMMARY:
This is a study to allow continued treatment for participants enrolled in studies of BXQ-350. This study is intended only for those who have completed the required study observation period or are still on treatment upon the closure of their respective BXQ-350 clinical study. The additional treatment is optional and voluntary.

DETAILED DESCRIPTION:
This is an open-label, multi-center, rollover study to allow continued treatment access for participants enrolled in studies of BXQ-350. This study is intended for subjects who have completed the required study observation period or are still on treatment upon the closure of their respective BXQ-350 clinical study, and who are judged by the Investigator to benefit from continued treatment with BXQ-350. The additional treatment is optional and voluntary.

This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.)

ELIGIBILITY:
Inclusion Criteria:

* Each subject must meet the following criteria:

  1. Has participated in and completed all protocol-specified treatments through the required study observation period or time of closure for a prior Bexion-sponsored BXQ-350 clinical study
  2. Has completed the End of Study visit of the prior Bexion-sponsored BXQ-350 clinical study
  3. Did not meet any treatment discontinuation criteria of the original prior Bexion- sponsored BXQ-350 clinical study
  4. Investigator opinion indicates that continued treatment with BXQ-350 is clinically appropriate for the subject
  5. Provide signed, written informed consent prior to the initiation of any study-specific procedures (Consent from Guardians for minor children and patient assent according to Institution and Institutional Review Board (IRB) standards)
  6. Have a negative serum pregnancy test result within 28 days prior to the first continuing treatment assessment for females of child bearing potential (FCBP); not applicable to subjects who are unable to become pregnant, including those with tubal ligation, bilateral oophorectomy and/or hysterectomy)
  7. FCBP and male subjects whose sexual partner(s) are FCBP must agree to abstain from heterosexual activity or use a double barrier method of contraception (e.g., condom and occlusive cap with spermicide) or highly effective contraception (intrauterine device or system, established hormonal contraceptive methods on a stable dose from the time of the last menstrual cycle, or vasectomized partner with confirmed azoospermia) from the time of study entry to 1 month after the last day of treatment

     Exclusion Criteria:
* Subjects must not meet any of the following criteria:

  1. Has any ongoing adverse event that could impact tolerability to BXQ-350
  2. Receiving any other non-BXQ-350 study treatment modalities with curative intent, including investigational products other than BXQ-350
  3. Are pregnant or nursing (lactating), where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive serum human chorionic gonadotropin (hCG) laboratory test

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with clinical benefit | Day 1 up to approximately 5 years
  Subjects will be assessed at every visit for continued clinical benefit as per Investigator's assessment.

SECONDARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events as Assessed by CTCAE v5.0 | Day 1 up to approximately 5 years
  Subjects will be assessed at every visit for adverse events
Time to Disease Progression | From Day 1 until the date of first documented disease progression or date of death from any cause, whichever occurs first; up to approximately 5 years
  Subjects will be assessed for disease progression throughout the study per institutional standard of care.
Overall Survival | From date of BXQ-350 treatment completion until time of death from any cause; up to approximately 5 years
  Subjects will be followed monthly for survival upon completion of BXQ-350 treatment.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky
  - University of Cincinnati Barrett Center, Cincinnati, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No